CLINICAL TRIAL: NCT03561610
Title: Impact of a Novel Form of Oral Nutritional Supplement Application in Cancer Patients With a High Risk for Malnutrition
Brief Title: Novel Form of Nutritional Supplementation in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ONOM
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Cancer; Malnutrition; Cachexia
Keywords: cancer cachexia; malnutrition; nutritional supplement; sip feed; nutritional risk
MeSH Terms: conditions — Neoplasms; Malnutrition; Cachexia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1 (Active Comparator): normal Nutrition + sip feed (covers individual energy and nutrient demands)
  Interventions: Dietary Supplement: sip feed
- Study group 2 (Experimental): normal Nutrition + gumdrops (covers individual energy and nutrient demands)
  Interventions: Dietary Supplement: gumdrops

INTERVENTIONS:
Dietary Supplement: sip feed — normal oral Nutrition + sip feed (Fresubin2.0®; covers individual energy and nutrient demands; high in protein)
  Arms: Study group 1
Dietary Supplement: gumdrops — normal oral Nutrition + gumdrops (Nutrimed®; covers individual energy and nutrient demands; high in protein)
  Arms: Study group 2

SUMMARY:
This study evaluates if a novel form of oral nutritional Supplement application in the form of gumdrops may serve as an alternative to common sip Feeds in cancer patients with high risk for malnutrition. Within this context the Impact of these two different supplements on General condition, Quality of life, muscle function, Body composition, Appetite and Nutrition Status are investigated. Patients are randomly allocated either to a study group with oral Supplementation in the form of sip feed or to a study Group receiving gumdrops for 4 weeks. After a washout period of 5-7 days study Groups are switched for another 4 week Intervention period.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with solid and hematological malignancies
* BMI < 20 kg/m² and/or NRS-2002 Score ≥ 3

Exclusion Criteria:

* pregnant or nursing women
* persons with psychiatric disorders with doubts about legal and cognitive capacity
* participation in nutritional Intervention Trials within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Compliance | 4 weeks
  compliance of nutritional supplement intake assessed by Medication Adherence Report Scale (MARS-D); Total score ranges from 0-10 with a higher score indicating better adherence
Tolerance of the form of oral supplementation | 4 weeks
  assessment of hedonic and sensoric estimation of oral supplements by questionnaire

SECONDARY OUTCOMES:
Body weight | 4 weeks
  Body weight assessed by bioelectrical impedance analysis (in kg)
Body composition | 4 weeks
  Skeletal muscle mass, Fat mass assessed by bioelectrical impedance analysis (in kg)
Physical function - Isometric muscle strength | 4 weeks
  Hand grip strength assessed by hand dynamometer (in kg)
Physical function - Lower limb strength | 4 weeks
  30 second sit-to-stand test (number of sit-to-stand cycles)
Physical function - Endurance | 4 weeks
  Six-minute-walk test (walking distance in m)
Patient-reported performance status | 4 weeks
  ECOG performance status/Karnofsky index
subjective Physical activity | 4 weeks
  Physical activity Level assessed by International Physical Activity Questionnaire (IPAQ)
objective Physical activity | 4 weeks
  Physical activity Level assessed by pedometer
Patient-reported Quality of Life (QoL) | 4 weeks
  EORTC QLQ - C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No